CLINICAL TRIAL: NCT04853823
Title: A Phase I, Single-Center, Double-Blind, Randomized Safety, Tolerability, and Dermal Reactogenicity Study of PDC-APB in Healthy Volunteers With a History of Contact Dermatitis Due to Poison Ivy Exposure
Brief Title: A Safety, Tolerability, and Dermal Reactogenicity Study of PDC-APB
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hapten Sciences, Inc. (Industry)
Collaborators: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PDC-APB CL-04
Record Dates: First submitted 2021-04-13; First posted 2021-04-21 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-04

CONDITIONS: Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Contact | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PDC-APB (Experimental): Study duration for each subject is approximately 15 weeks (105 days) for Screening including patch testing, Treatment, and the initial 30-day post-treatment periods. Approximately 6 weeks after treatment, subjects will receive a second patch test. In addition, each subject will be followed from T1 for 6 months by monthly telephone follow-up to monitor adverse events. Subjects in Cohorts 2, 3 and 4 and, if applicable, additional cohorts, will not be dosed until all subjects from the prior cohort have completed the assessments after IP dosing and the Safety Review Committee has reviewed the results prior to Day T14. All subjects will be followed for 6 months after IP dosing for safety assessments, which will be carried out at monthly intervals via telephone.
  Interventions: Drug: PDC-APB
- Vehicle (Placebo Comparator): Study duration for each subject is approximately 15 weeks (105 days) for Screening including patch testing, Treatment, and the initial 30-day post-treatment periods. Approximately 6 weeks after treatment, subjects will receive a second patch test. In addition, each subject will be followed from T1 for 6 months by monthly telephone follow-up to monitor adverse events. Subjects in Cohorts 2, 3 and 4 and, if applicable, additional cohorts, will not be dosed until all subjects from the prior cohort have completed the assessments after IP dosing and the Safety Review Committee has reviewed the results prior to Day T14. All subjects will be followed for 6 months after IP dosing for safety assessments, which will be carried out at monthly intervals via telephone.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PDC-APB — PDC-APB Intra-muscular Injection
  Other Names: Active
  Arms: PDC-APB
Other: Placebo — Vehicle
  Other Names: Vehicle
  Arms: Vehicle

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose study to assess the safety and tolerability of PDC-APB by intramuscular (IM) injection compared to placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single ascending dose study to assess the safety, tolerability and dermal reactogenicity in subjects shown to be sensitive to urushiol of PDC-APB by intramuscular (IM) injection compared to placebo. In this study, it is anticipated that up to 4 dose levels (5.0 mg, 10 mg, 15 mg, and 20 mg PDC-APB) will be studied in sequential cohorts. Each cohort will enroll 8 subjects, 6 subjects randomized to active treatment and 2 randomized to placebo, in a double-blind manner.

Safety will be assessed in each cohort before starting treatment at the next higher dose level. If the study treatment is tolerated and there are no findings that necessitate stopping the study, the next cohort will be treated at the next higher dose level, in the same manner. This process will continue until the highest intended dose is reached, or side effects that limit further dose escalation are observed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects, as determined by medical history and physical examination, from 18 to 65 years of age, inclusive.
2. Documented history of urushiol exposure on the Allergic Contact Dermatitis Questionnaire.
3. For female subjects: Surgically sterile or menopausal (at least 1-year absence of vaginal bleeding or spotting). Females of childbearing age/potential may be included provided they are using medically acceptable methods of birth control for 1 month prior to and for the duration of the study and 3 months thereafter. Dual methods, for example, a hormonal method used with a barrier method, must be used.
4. For male subjects and their partners of childbearing potential: Willing to use 2 methods of contraception, 1 of which must be a barrier method, for the duration of the study and 3 months after the last dose of IP, and agree to not donate sperm for 3 months after the last dose of IP.
5. Has sufficient normal skin area on the back to accommodate two patch applications (no scarring, acne, excessive hair, or tattooing)
6. Able to participate and willing to give written informed consent and to comply with the study restrictions.

Exclusion Criteria:

1. History of alcohol or drug abuse within the past 24 months or related concerns of the investigator.
2. Positive human immunodeficiency (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) clinical laboratory test.
3. Administration of, or need for, any prescription drug within 30 days, or over-the-counter (OTC) drugs on a regular basis. Hormonal contraceptive drugs, hormone replacement therapy (stable dose for at least 3 months), acetaminophen and ibuprofen ≤ 1 g/day, blood pressure and cholesterol medication, anti-acids, and multivitamins are permitted.
4. Any screening laboratory evaluation for liver function outside the laboratory reference range or any other laboratory value > 1.5 × the reference range not approved in writing by the Medical Monitor.
5. Body temperature > 37.5°C (99.5°F), systolic blood pressure (SBP) < 90 or > 139 mmHg, diastolic blood pressure (DBP) < 50 or > 89 mmHg, or presence of any other abnormal vital signs measurement considered by the Investigator to be clinically significant.
6. History of clinically significant renal or urinary disease or active symptoms of renal or urinary disease. A history of renal stones or urinary tract infections does not exclude a subject.
7. History of clinically significant hepatic disease or impairment, or any active symptoms of hepatic disease.
8. Presence of clinically significant gastrointestinal (GI) disorder or symptoms of active GI disease. A history of appendectomy or cholecystectomy does not exclude a subject.
9. History of significant cardiovascular disease, congestive heart failure, stroke, angina, arrhythmias, or symptoms or signs of active cardiovascular disease, or a clinically significant abnormality on the screening ECG considered by the Sponsor and the Investigator to be unacceptable. Hypertension and hypercholesterolemia if well-controlled are not excluded.
10. History of clinically significant psychiatric disease, including but not limited to bipolar disorder, depression, anxiety, panic attacks, and schizophrenia.
11. History or symptoms of clinically significant central nervous system disease, including but not limited to transient ischemic attack, stroke, seizure disorder, history of loss of consciousness or head trauma, or behavioral disturbances.
12. History of suicide attempt or report of suicidal ideation.
13. Concomitant disease or any organ system condition or abnormality that could pose an unacceptable risk to the subject in this study, in the opinion of the Investigator, based on possible interference with absorption, distribution, metabolism, or elimination of the IP or possible effect of the IP on the condition or abnormality.
14. History of clinically significant allergies requiring treatment with steroids (by topical or oral administration) in the previous 90 days, use in the previous year of any immunosuppressants or immunotherapy, or use of oral or topical antihistamines in the previous 30 days.
15. Known or suspected allergy or cutaneous sensitivity to any product components, including sesame or sesame oil, benzyl alcohol, or ethanol.
16. History of asthma, including subjects with asthma who require acute or maintenance inhaled or oral steroid use for control of symptoms, as well as subjects with intermittent asthma who do not require corticosteroids.
17. History of any acute or chronic skin condition (except acne or contact dermatitis as noted in Inclusion Criteria #2) or the presence of any rashes on the back at screening or baseline that would interfere with patch assessments.
18. Presence of tattoos or skin disease at the intended patch application sites.
19. Participation in an investigational drug or device study within 30 days prior to screening.
20. Unwillingness or inability to comply with the study protocol for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events [Safety and tolerability] | 24 Weeks
  The Primary outcome measure for this study will be the overall safety profile observed during the post-treatment observation period in the study population. AEs will be classified by organ class using the coding system and by severity (Grades 1-4, Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials).
  The primary objective of the study is to assess the safety and tolerability of PDC-APB following single doses administered intramuscularly to healthy subjects between 18 and 65 years of age.

SECONDARY OUTCOMES:
Urushiol Sensitivity [scored +/-, 0-4] | 15 Weeks
  Secondary assessments will evaluate the effect of PDC-APB injection on urushiol sensitivity (scored +/-, 0-4). Local reactogenicity to the second urushiol patch applied 6 weeks after IP injection will be compared to the reactogenicity scores following application of the first patch 6 weeks prior to injection of IP.

CONTACTS AND LOCATIONS:
Overall Officials: James Marks, MD, Principal Investigator — Milton S. Hershey Medical Center

IPD SHARING:
Plan to Share IPD: No